CLINICAL TRIAL: NCT06633770
Title: Role of Presepsin as a Novel Biomarker in Diagnosis of Neonatal Sepsis
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sara Saleh Ahmed, resident-clinical pathology sohag university hospital, Sohag University
Other Study IDs: soh-Med-24-09-11MS
Record Dates: First submitted 2024-10-02; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Neonatal Sepsis
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- (case group):: Consists of 70 neonates, whose blood culture results were positive and indicative of known sepsis-causing pathogens and neonates whose clinical and laboratory findings were indicative of probable sepsis despite negative blood culture results.
  Clinical and laboratory findings were indicative of probable sepsis :
  * Fever or low temperature.
  * Fast or slow heart rate.
  * Fast breathing or shortness of breath.
  * Vomiting.
  * Diarrhea.
  * Reduced sucking/difficulty feeding.
  * Swollen belly (abdomen).
  * Cold hands and feet.
  * Leukocyte (<5000 or ≥20000 wbcs/ µL), absolute neutrophil (>60%) a
  * Thrombocytopenia:
  Interventions: Diagnostic Test: proclcitonin and presepsin
- control group: 30 healthy neonates who had no signs of sepsis in clinical, radiographic, or laboratory findings or whose symptoms could be characteristic of another disease.
  Interventions: Diagnostic Test: proclcitonin and presepsin

INTERVENTIONS:
Diagnostic Test: proclcitonin and presepsin — All included patients will be subjected to:
  * laboratory investigations
    * Complete Blood Count (CBC),
    * Liver Function Test(LFT) ( ALT,AST, Billirubin, total protein and albumin)
    * Kidney function test (KFT) ( Urea and creatinine)
    * Random Blood Glucose (RBG).
    * Erythrocyte Sedimentation Rate(ESR )
    * Urine analysis -A special investigations include (blood culture, C Reactive protein (CRP), proclcitonin and presepsin).

SUMMARY:
-Introduction: Sepsis is a clinical syndrome that results from a deregulated inflammatory response to an infection. it is life-threatening entity causing millions of deaths worldwide, with variable clinical manifestations and poses difficulty in diagnosis and treatment. Early recognition of sepsis not only helps in the optimization of treatment but also improves the overall outcome.

Neonatal sepsis is generally considered a spectrum of disorders that result from infection by bacteria , viruses, fungi ,or parasites or the toxic products of these., It is characterized by nonspecific signs and symptoms so it is a conundrum of diagnostic and therapeutic challenges .The proof of infection is seldom encountered in practice, as the confirmatory microbial culture yield can be as low as 25-30%. Hence, clinicians often depend on commonly available biomarkers such as C-reactive Protein (CRP) and procalcitonin (PCT) for diagnosing infection. Even though helpful, these markers are fraught with errors and limitations There is an exigent need for a novel biomarker that can serve as a clear distinguisher of sepsis from other non-septic inflammatory conditions The role of presepsin as a biomarker of sepsis in children is still a matter of scientific inquiry.

CD14 is a co-receptor present on the surface of the monocyte/macrophage. It is a member of the Toll-like receptors (TLRs),with an ability to identify groups of ligands of both gram-positive and gram-negative pathogens CD14 exists in two forms namely membrane-bound (mCD14) and a soluble form (sCD14). The sCD14 has different subtypes that get released in circulation and acted upon by proteases and cathepsin D . The N terminal fragment of the sCD14-ST subtype is called presepsin.

ELIGIBILITY:
Inclusion Criteria:

* Neonates from 0 to 1 month of age of both sexes included in this study with any suspected case of neonatal sepsis with maternal risk factors for sepsis, e.g., ( prolonged labor, premature rupture of membrane (PROM), maternal intrapartum fever and chorioamnionitis,) and neonates with sepsis-related clinical signs: (temperature instability, apnea, need for supplemental oxygen, bradycardia, tachycardia, hypotension, hypoperfusion, feeding intolerance, and abdominal distension).

Exclusion Criteria:

* Administration of antibiotic therapy prior to admission, Birth asphyxia Laboratory finding suggestive of inborn error of metabolism Congenital anomalies including congenital heart disease

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Neonates from 0 to 1 month of age of both sexes included in this study with any suspected case of neonatal sepsis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
• The outcomes of interest for the analyses were presepsin sensitivity, specificity, and diagnostic odds ratio for the diagnosis of neonatal sepsis | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Strunk T, Molloy EJ, Mishra A, Bhutta ZA. Neonatal bacterial sepsis. Lancet. 2024 Jul 20;404(10449):277-293. doi: 10.1016/S0140-6736(24)00495-1. Epub 2024 Jun 26. PMID 38944044
- [Background] Pospisilova I, Brodska HL, Bloomfield M, Borecka K, Janota J. Evaluation of presepsin as a diagnostic tool in newborns with risk of early-onset neonatal sepsis. Front Pediatr. 2023 Jan 9;10:1019825. doi: 10.3389/fped.2022.1019825. eCollection 2022. PMID 36699313
- [Background] Wei S, Shen Z, Yin Y, Cong Z, Zeng Z, Zhu X. Advances of presepsin in sepsis-associated ARDS. Postgrad Med J. 2024 Mar 18;100(1182):209-218. doi: 10.1093/postmj/qgad132. PMID 38147883
- [Background] Krack AT, Eckerle M, Mahajan P, Ramilo O, VanBuren JM, Banks RK, Casper TC, Schnadower D, Kuppermann N; Febrile Infant Working Group of the Pediatric Emergency Care Applied Research Network (PECARN). Leukopenia, neutropenia, and procalcitonin levels in young febrile infants with invasive bacterial infections. Acad Emerg Med. 2024 Sep;31(9):903-914. doi: 10.1111/acem.14921. Epub 2024 Apr 25. PMID 38661246
- [Background] Poggi C, Lucenteforte E, Petri D, De Masi S, Dani C. Presepsin for the Diagnosis of Neonatal Early-Onset Sepsis: A Systematic Review and Meta-analysis. JAMA Pediatr. 2022 Aug 1;176(8):750-758. doi: 10.1001/jamapediatrics.2022.1647. PMID 35639395